CLINICAL TRIAL: NCT01678924
Title: A Safety and Efficacy Study of AGN-214868 in Patients With Postherpetic Neuralgia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 214868-007; 2012-002240-24 (EudraCT Number)
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Results first posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Neuralgia, Postherpetic
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- AGN-214868 Dose 1 (Experimental): AGN-214868 Dose 1 given as injections into the area of pain on Day 1.
  Interventions: Drug: AGN-214868
- AGN-214868 Dose 2 (Experimental): AGN-214868 Dose 2 given as injections into the area of pain on Day 1.
  Interventions: Drug: AGN-214868
- AGN-214868 Placebo (Vehicle) (Placebo Comparator): AGN-214868 placebo (vehicle) given as injections into the area of pain on Day 1.
  Interventions: Drug: AGN-214868 Placebo (Vehicle)
- AGN-214868 Dose 3 (Experimental): AGN-214868 Dose 3 given as injections into the area of pain on Day 1.
  Interventions: Drug: AGN-214868

INTERVENTIONS:
Drug: AGN-214868 — AGN-214868 given as injections into the area of pain on Day 1.
  Arms: AGN-214868 Dose 1; AGN-214868 Dose 2; AGN-214868 Dose 3
Drug: AGN-214868 Placebo (Vehicle) — AGN-214868 placebo (vehicle) given as injections into the area of pain on Day 1.
  Arms: AGN-214868 Placebo (Vehicle)

SUMMARY:
This is a safety and efficacy study of AGN-214868 in patients with postherpetic neuralgia (PHN).

ELIGIBILITY:
Inclusion Criteria:

* Postherpetic neuralgia with pain present for at least 9 months

Exclusion Criteria:

* Active herpes zoster skin rash
* Anticipated treatment for postherpetic neuralgia during the first 3 months of the study, including oral and topical medications, acupuncture, spinal cord stimulation, transcutaneous nerve stimulation (TNS), or trigger point injection
* Anticipated treatment with pain medication for the treatment of postherpetic neuralgia during the first 3 months of the study
* Use of capsaicin treatment for postherpetic neuralgia within 6 months, or anticipated use during the first 3 months of the study
* Use of botulinum toxin of any serotype for any reason within 6 months, or anticipated use during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (69):
- United States (33):
  - Agave Clinical Research, LLC, Mesa, Arizona
  - Territory Neurology & Research Institute, Tucson, Arizona
  - Neuro-Pain Medical Center, Fresno, California
  - University of California, Irvine, Irvine, California
  - Loma Linda University, Loma Linda, California
  - Northern California Research Corp, Sacramento, California
  - Neurological Research Institute, Santa Monica, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - The Mile High Research Center, Denver, Colorado
  - Riverside Clinical Research, Edgewater, Florida
  - Compass Research, LLC, Orlando, Florida
  - Drug Studies America, Marietta, Georgia
  - Injury Care Research, LLC, Boise, Idaho
  - Millennium Pain Center, Bloomington, Illinois
  - Beacon Clinical Research, Brockton, Massachusetts
  - Springfield Neurology Associates, LLC, Springfield, Massachusetts
  - Michigan Head Pain and Neurology Institute, Ann Arbor, Michigan
  - Quest Research Institute, Farmington Hills, Michigan
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Clinvest Headache Care Center, Springfield, Missouri
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - The Medical Research Network, LLC, New York, New York
  - Island Neurological Associates, P.C., Plainview, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Plains Medical Clinic, Fargo, North Dakota
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - Allegheny Pain Management, Altoona, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Clinical Trials of South Carolina, LLC, Charleston, South Carolina
  - PharmaCorp Clinical Trials, Inc, Charleston, South Carolina
  - Clinical Research of Charleston, Mt. Pleasant, South Carolina
  - Center for Clinical Studies, Webster, Texas
  - MultiCare Neuroscience Center of Washington, Tacoma, Washington
- Austria (3):
  - AKH Wien, Vienna
  - Wilhelminenspital der Stadt Wien, Vienna
  - SMZ-Ost Donauspital, Vienna
- Germany (21):
  - Pro scientia med im MARE Klinikum, Kiel, Schleswig-Holstein
  - Berlin Research Centre, Berlin
  - Regionales Schmerzzentrum DGS, Bielefeld
  - Bochum Research Centre, Bochum
  - Das Schmerzzentrum Celle, Celle
  - Ambulant study centre, Cologne
  - Leiter des Universitats Schmerz Centrums (USC), Dresden
  - Neuro-Consil GmbH, Düsseldorf
  - Frankfurt Research Centre, Frankfurt
  - Schmerz und Palliativzentrum Fulda, Fulda
  - Schmerz und Palliativ- Zentrum Goeppingen, Göppingen
  - Klinikum Hanau GmbH, Hanau
  - Neurologische Praxis Heidenheim, Heidenheim
  - Facharzt fur Neurologie, Hoppegarten
  - Schmerzklinik Kiel, Kiel
  - Medamed GmbH, Leipzig
  - Leipzig Research Centre, Leipzig
  - Magdeburg Research Centre, Magdeburg
  - Regionales Schmerz- und Palliativ Zentrum DGS Mainz, Mainz
  - Universitätsklinik Ulm, Ulm
  - Schmerztherapiezentrum Villingen-Schwenningen, Villingen-Schwenningen
- Poland (12):
  - Poznański Ośrodek Medyczny NOVAMED, Poznan, Poznañ
  - Medica Pro Familia Sp. Z.o.o SKA, Gdynia
  - Medica Pro Familia Sp. Z.o.o SKA, Katowice
  - Malopolskie Centrum Medyczne S.C., Krakow
  - Specjalistyczny Gabinet Neurologiczny, Krakow
  - Nzoz Neuromed, Lublin
  - NZOZ Neuro-Kard, Poznan
  - Osrodek Badan Klinicznych Euromedis Sp. z o.o., Szczecin
  - Niepubliczny Zaklad Opieki Zdrowotnej, Świdnik
  - Przychodnia Specjalistyczna PROSEN, Warsaw
  - Medica Pro Familia Warszawa, Warsaw
  - Synexus SCM sp. z o.o., Wroclaw

RESULTS

PARTICIPANT FLOW:
Groups:
- AGN 214868 130µg; AGN 214868 65µg; AGN 214868 32.5µg: Single administration of AGN-214868, total dose given as injections into the area of pain on Day 1
- Placebo: Single administration of AGN-214868 placebo, given as injections into the area of pain on Day 1
Period: Overall Study
Arm/Group | AGN 214868 130µg | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Started | 64 | 63 | 30 | 123
Completed | 54 | 51 | 28 | 105
Not Completed | 10 | 12 | 2 | 18
Not completed — Adverse Event | 1 | 1 | 0 | 1
Not completed — Lack of Efficacy | 7 | 2 | 0 | 5
Not completed — Lost to Follow-up | 0 | 4 | 0 | 2
Not completed — Personal Reasons | 2 | 2 | 2 | 7
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 2
Not completed — Unable to attend scheduled visits | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population, consisting of patients who received 1 dose of study drug in the study, included 280 patients
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN 214868 130µg | AGN 214868 65µg | AGN 214868 32.5µg | Placebo | Total
Number analyzed (Participants) | 64 | 63 | 30 | 123 | 280
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (10.47) | 65.3 (12.82) | 65.0 (11.99) | 67.0 (8.13) | 66.3 (10.28)
Age, Customized [Number; unit: participants]
  18 years to less than 40 years | 1 | 3 | 1 | 0 | 5
  40 years to less than 65 years | 20 | 19 | 12 | 46 | 97
  65 years and over | 43 | 41 | 17 | 77 | 178
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 37 | 34 | 13 | 50 | 134
  Female | 27 | 29 | 17 | 73 | 146
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 56 | 52 | 26 | 112 | 246
  Black | 3 | 4 | 1 | 7 | 15
  Asian | 0 | 2 | 2 | 1 | 5
  Hispanic | 5 | 4 | 1 | 2 | 12
  Other | 0 | 1 | 0 | 1 | 2
Weight [Mean (Standard Deviation); unit: kg] | 84.9 (19.15) | 82.3 (17.67) | 80.0 (14.48) | 78.8 (17.83) | 81.1 (17.86)
Height [Mean (Standard Deviation); unit: cm] | 169.8 (10.22) | 167.7 (10.98) | 169.1 (8.91) | 166.4 (9.07) | 167.7 (9.83)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Pain Intensity Score - Cohort 1
Description: The average pain intensity score at each week was the mean of the daily average pain intensity scores reported in the patient's eDiary during each 7-day period, starting with the day of study treatment injection. Patients used the 11-point Likert scale, with anchors at 0 = "no pain" and 10 = "pain as bad as you can imagine" Baseline was defined as the mean of the daily average pain intensity scores reported during the baseline period for the 7 days immediately prior to the treatment.
Time Frame: Baseline to Week 12
Population: Two cohorts of patients with postherpetic neuralgia (PHN) were randomized to receive 1 treatment of either AGN-214868 (cohort 1: 32.5 or 65 μg; cohort 2: 130 μg) or placebo. Cohort 1 includes 154 patients from the modified intent to treat (mITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 63 | 30 | 61
units on a scale
  Week 1 | -0.88 [-1.249 to -0.538] | -1.02 [-1.380 to -0.587] | -1.11 [-1.425 to -0.808]
  Week 2 | -1.33 [-1.746 to -0.968] | -1.56 [-1.963 to -1.017] | -1.57 [-1.970 to -1.174]
  Week 3 | -1.66 [-2.143 to -1.203] | -1.93 [-2.426 to -1.227] | -1.84 [-2.248 to -1.388]
  Week 4 | -1.78 [-2.277 to -1.310] | -2.20 [-2.721 to -1.432] | -1.98 [-2.423 to -1.482]
  Week 5 | -1.83 [-2.321 to -1.384] | -2.19 [-2.675 to -1.379] | -2.10 [-2.557 to -1.554]
  Week 6 | -1.97 [-2.442 to -1.495] | -2.07 [-2.597 to -1.297] | -2.34 [-2.755 to -1.697]
  Week 7 | -2.00 [-2.481 to -1.506] | -2.08 [-2.572 to -1.328] | -2.32 [-2.746 to -1.673]
  Week 8 | -2.11 [-2.591 to -1.618] | -2.02 [-2.530 to -1.263] | -2.40 [-2.825 to -1.745]
  Week 9 | -2.21 [-2.66 to -1.701] | -2.15 [-2.682 to -1.352] | -2.52 [-2.805 to -1.733]
  Week 10 | -2.28 [-2.679 to -1.674] | -2.29 [-2.812 to -1.481] | -2.48 [-2.743 to -1.634]
  Week 11 | -2.27 [-2.684 to -1.672] | -2.46 [-2.996 to -1.570] | -2.56 [-2.807 to -1.724]
  Week 12 | -2.20 [-2.626 to -1.600] | -2.53 [-3.061 to -1.605] | -2.65 [-2.886 to -1.783]

2. Primary Outcome: Change From Baseline in Average Pain Intensity Score - Cohort 2
Description: as for outcome 1
Time Frame: Baseline to Week 12
Population: Two cohorts of patients with postherpetic neuralgia (PHN) were randomized to receive 1 treatment of either AGN-214868 (cohort 1: 32.5 or 65 μg; cohort 2: 130 μg) or placebo. Cohort 2 includes 125 patients from the mITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 64 | 61
units on a scale
  Week 1 | -0.78 [-1.093 to -0.451] | -0.88 [-1.190 to -0.492]
  Week 2 | -1.12 [-1.508 to -0.701] | -1.37 [-1.791 to -0.799]
  Week 3 | -1.45 [-1.788 to -0.952] | -1.65 [-2.064 to -1.057]
  Week 4 | -1.62 [-1.934 to -1.072] | -1.90 [-2.344 to -1.269]
  Week 5 | -1.88 [-2.202 to -1.301] | -1.88 [-2.366 to -1.257]
  Week 6 | -2.04 [-2.226 to -1.305] | -1.90 [-2.339 to -1.235]
  Week 7 | -2.14 [-2.345 to -1.352] | -1.90 [-2.352 to -1.225]
  Week 8 | -2.29 [-2.405 to -1.404] | -1.96 [-2.412 to -1.270]
  Week 9 | -2.35 [-2.493 to -1.497] | -2.00 [-2.457 to -1.293]
  Week 10 | -2.44 [-2.584 to -1.557] | -2.04 [-2.515 to -1.311]
  Week 11 | -2.49 [-2.647 to -1.581] | -2.03 [-2.489 to -1.314]
  Week 12 | -2.49 [-2.659 to -1.632] | -2.03 [-2.538 to -1.354]

3. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 1 - Week 1
Description: Average Pain Intensity Score Responder is defined as a patient who had at least a 30% improvement (decrease) in average pain intensity score at each week compared with baseline
Time Frame: Baseline to Week 1
Population: The total modified intent to treat (mITT) population of 279 patients, consists of all randomized patients who received treatment and at least 1 post-baseline weekly average pain intensity score. Cohort 1 includes 154 patients from the mITT population
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 61 | 30 | 61
percentage of patients | 18.0 | 33.3 | 21.3

4. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 1 - Week 2
Description: as for outcome 3
Time Frame: Baseline to Week 2
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 63 | 30 | 60
percentage of patients | 27.0 | 40.0 | 36.7

5. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 1 - Week 3
Description: as for outcome 3
Time Frame: Baseline to Week 3
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 60 | 30 | 60
percentage of patients | 35.0 | 50.0 | 50.0

6. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 1 - Week 4
Description: Average Pain Intensity Score Responder is defined as a patient who had at least a 30% improvement (decrease), and in 10% increments, up to 100% improvement, in average pain intensity score at each week compared with baseline
Time Frame: Baseline to Week 4
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 61 | 30 | 59
percentage of patients | 37.7 | 53.3 | 50.8

7. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 1 - Week 5
Description: as for outcome 3
Time Frame: Baseline to Week 5
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 59 | 30 | 57
percentage of patients | 40.7 | 53.3 | 52.6

8. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 1 - Week 6
Description: as for outcome 3
Time Frame: Baseline to Week 6
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 58 | 30 | 55
percentage of patients | 41.4 | 50.0 | 54.5

9. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 1 - Week 7
Description: as for outcome 3
Time Frame: Baseline to Week 7
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 60 | 30 | 57
percentage of patients | 43.3 | 56.7 | 50.9

10. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 1 - Week 8
Description: as for outcome 3
Time Frame: Baseline to Week 8
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 58 | 30 | 56
percentage of patients | 43.1 | 50.0 | 55.4

11. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 1 - Week 9
Description: as for outcome 3
Time Frame: Baseline to Week 9
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 55 | 27 | 52
percentage of patients | 43.6 | 51.9 | 51.9

12. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 1 - Week 10
Description: as for outcome 3
Time Frame: Baseline to Week 10
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 56 | 28 | 52
percentage of patients | 46.4 | 53.6 | 55.8

13. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 1 - Week 11
Description: as for outcome 3
Time Frame: Baseline to Week 11
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 53 | 28 | 52
percentage of patients | 47.2 | 53.6 | 59.6

14. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 1 - Week 12
Description: as for outcome 3
Time Frame: Baseline to Week 12
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 50 | 27 | 49
percentage of patients | 48.0 | 63.0 | 63.3

15. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 2 - Week 1
Description: as for outcome 3
Time Frame: Baseline to Week 1
Population: The total mITT population of 279 patients, consists of all randomized patients who received treatment and at least 1 post-baseline weekly average pain intensity score. The mITT population for Cohort 2 is 125 patients
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 63 | 59
percentage of patients | 14.3 | 20.3

16. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 2 - Week 2
Description: as for outcome 3
Time Frame: Baseline to Week 2
Population: as for outcome 15
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 62 | 58
percentage of patients | 25.8 | 27.6

17. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 2 - Week 3
Description: as for outcome 3
Time Frame: Baseline to Week 3
Population: as for outcome 15
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 59 | 58
percentage of patients | 30.5 | 39.7

18. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 2 - Week 4
Description: as for outcome 3
Time Frame: Baseline to Week 4
Population: as for outcome 15
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 60 | 58
percentage of patients | 35.0 | 43.1

19. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 2 - Week 5
Description: as for outcome 3
Time Frame: Baseline to Week 5
Population: as for outcome 15
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 57 | 57
percentage of patients | 42.1 | 45.6

20. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 2 - Week 6
Description: as for outcome 3
Time Frame: Baseline to Week 6
Population: as for outcome 15
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 53 | 57
percentage of patients | 45.3 | 45.6

21. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 2 - Week 7
Description: as for outcome 3
Time Frame: Baseline to Week 7
Population: as for outcome 15
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 50 | 56
percentage of patients | 50.0 | 48.2

22. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 2 - Week 8
Description: as for outcome 3
Time Frame: Baseline to Week 8
Population: as for outcome 15
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 51 | 55
percentage of patients | 54.9 | 49.1

23. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 2 - Week 9
Description: as for outcome 3
Time Frame: Baseline to Week 9
Population: as for outcome 15
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 51 | 55
percentage of patients | 58.8 | 45.5

24. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 2 - Week 10
Description: as for outcome 3
Time Frame: Baseline to Week 10
Population: as for outcome 15
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 51 | 55
percentage of patients | 64.7 | 47.3

25. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 2 - Week 11
Description: as for outcome 3
Time Frame: Baseline to Week 11
Population: as for outcome 15
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 50 | 54
percentage of patients | 64.0 | 42.6

26. Secondary Outcome: Percentage of Average Pain Intensity Score Responders - Cohort 2 - Week 12
Description: as for outcome 3
Time Frame: Baseline to Week 12
Population: as for outcome 15
Measure: Number; unit: percentage of patients
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 44 | 50
percentage of patients | 61.4 | 40.0

27. Secondary Outcome: Change From Baseline in Maximal Area of Spontaneous Pain - Cohort 1 - Week 2
Description: The assessment of maximal area of spontaneous pain (MASP) was conducted by a qualified and trained investigator or designee (eg, physician, physician's assistant, nurse practitioner, and nurse). This assessment is based on color photographs taken of the patient and that the patient was asked to circle their MASP on with a black marker. Areas of pain were quantified at a central reading center.
Time Frame: Baseline to Week 2
Population: The total modified intent to treat (mITT) population of 279 patients, consists of all randomized patients who received treatment and at least 1 post-baseline weekly average pain intensity score assessment. Cohort 1 includes 154 patients from the mITT population
Measure: Least Squares Mean (95% Confidence Interval); unit: Square Centimeters (cm^2)
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 61 | 27 | 60
Square Centimeters (cm^2) | -25.07 [-37.544 to -13.564] | -34.07 [-60.871 to -4.114] | -26.10 [-38.580 to -14.053]

28. Secondary Outcome: Change From Baseline in Maximal Area of Spontaneous Pain - Cohort 1 - Week 4
Description: The assessment of maximal area of spontaneous pain (MASP) was conducted by a qualified and trained investigator or designee (eg, physician, physician's assistant, nurse practitioner, and nurse). This assessment is based on color photographs taken of the patient in which the patient was asked to outline their MASP with a black marker. Areas of pain were quantified at a central reading center.
Time Frame: Baseline to Week 4
Population: as for outcome 27
Measure: Least Squares Mean (95% Confidence Interval); unit: Square Centimeters (cm^2)
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 62 | 29 | 60
Square Centimeters (cm^2) | -27.65 [-40.978 to -15.412] | -25.96 [-49.316 to 0.309] | -32.23 [-48.543 to -16.214]

29. Secondary Outcome: Change From Baseline in Maximal Area of Spontaneous Pain - Cohort 1 - Week 8
Description: as for outcome 28
Time Frame: Baseline to Week 8
Population: as for outcome 27
Measure: Least Squares Mean (95% Confidence Interval); unit: Square Centimeters (cm^2)
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 56 | 28 | 55
Square Centimeters (cm^2) | -29.86 [-45.876 to -15.566] | -37.18 [-64.825 to -1.989] | -34.04 [-48.026 to -22.134]

30. Secondary Outcome: Change From Baseline in Maximal Area of Spontaneous Pain - Cohort 1 - Week 12
Description: as for outcome 28
Time Frame: Baseline to Week 12
Population: as for outcome 27
Measure: Least Squares Mean (95% Confidence Interval); unit: Square Centimeters (cm^2)
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 57 | 29 | 54
Square Centimeters (cm^2) | -30.99 [-46.118 to -17.138] | -31.40 [-61.185 to 3.853] | -35.03 [-53.242 to -18.425]

31. Secondary Outcome: Change From Baseline in Maximal Area of Spontaneous Pain - Cohort 2 - Week 2
Description: as for outcome 28
Time Frame: Baseline to Week 2
Population: The total mITT population of 279 patients, consists of all randomized patients who received treatment and at least 1 post-baseline weekly average pain intensity score assessment. The mITT population for Cohort 2 is 125 patients
Measure: Least Squares Mean (95% Confidence Interval); unit: Square Centimeters (cm^2)
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 57 | 57
Square Centimeters (cm^2) | -9.86 [-38.087 to 18.020] | -27.52 [-43.841 to -10.854]

32. Secondary Outcome: Change From Baseline in Maximal Area of Spontaneous Pain - Cohort 2 - Week 4
Description: as for outcome 28
Time Frame: Baseline to Week 4
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: Square Centimeters (cm^2)
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 58 | 59
Square Centimeters (cm^2) | -22.23 [-48.893 to 3.903] | -25.67 [-42.901 to -7.909]

33. Secondary Outcome: Change From Baseline in Maximal Area of Spontaneous Pain - Cohort 2 - Week 8
Description: as for outcome 28
Time Frame: Baseline to Week 8
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: Square Centimeters (cm^2)
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 53 | 57
Square Centimeters (cm^2) | -42.92 [-65.580 to -23.080] | -31.95 [-47.299 to -13.978]

34. Secondary Outcome: Change From Baseline in Maximal Area of Spontaneous Pain - Cohort 2 - Week 12
Description: as for outcome 28
Time Frame: Baseline to Week 12
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: Square Centimeters (cm^2)
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 54 | 57
Square Centimeters (cm^2) | -36.73 [-67.719 to -8.696] | -32.60 [-49.823 to -12.574]

35. Secondary Outcome: Change From Baseline in Area of Allodynia - Cohort 1 - Week 2
Description: The assessment of maximal area of allodynia was conducted by a qualified and trained investigator or designee (eg, physician, physician's assistant, nurse practitioner, and nurse). This assessment is based on color photographs taken of the patient in which the patient was asked to outline their maximal area of skin that feels unpleasant to the touch (allodynic skin) with a red marker. Areas of allodynia were quantified at a central reading center.
Time Frame: Baseline to Week 2
Population: The total mITT population of 279 patients, consists of all randomized patients who received treatment and at least 1 post-baseline weekly average pain intensity score assessment. The mITT population for Cohort 1 is 154 patients.
Measure: Least Squares Mean (95% Confidence Interval); unit: Square Centimeters (cm^2)
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 61 | 27 | 60
Square Centimeters (cm^2) | -40.06 [-89.750 to -12.158] | -14.42 [-34.431 to 23.824] | -52.73 [-67.258 to -24.248]

36. Secondary Outcome: Change From Baseline in Area of Allodynia - Cohort 1 - Week 4
Description: as for outcome 35
Time Frame: Baseline to Week 4
Population: as for outcome 35
Measure: Least Squares Mean (95% Confidence Interval); unit: Square Centimeters (cm^2)
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 62 | 29 | 60
Square Centimeters (cm^2) | -54.12 [-118.867 to -19.566] | -23.07 [-41.985 to 19.468] | -58.14 [-70.452 to -26.048]

37. Secondary Outcome: Change From Baseline in Area of Allodynia - Cohort 1 - Week 8
Description: as for outcome 35
Time Frame: Baseline to Week 8
Population: as for outcome 35
Measure: Least Squares Mean (95% Confidence Interval); unit: Square Centimeters (cm^2)
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 56 | 28 | 55
Square Centimeters (cm^2) | -74.46 [-136.541 to -43.526] | -50.47 [-75.433 to -4.124] | -71.54 [-85.155 to -37.104]

38. Secondary Outcome: Change From Baseline in Area of Allodynia - Cohort 1 - Week 12
Description: as for outcome 35
Time Frame: Baseline to Week 12
Population: as for outcome 35
Measure: Least Squares Mean (95% Confidence Interval); unit: Square Centimeters (cm^2)
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 57 | 29 | 54
Square Centimeters (cm^2) | -67.71 [-130.695 to -35.611] | -39.96 [-62.646 to 8.446] | -70.46 [-92.167 to -29.970]

39. Secondary Outcome: Change From Baseline in Area of Allodynia - Cohort 2 - Week 2
Description: as for outcome 35
Time Frame: Baseline to Week 2
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: Square Centimeters (cm^2)
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 57 | 57
Square Centimeters (cm^2) | -36.66 [-59.461 to -0.328] | -60.71 [-98.564 to -36.369]

40. Secondary Outcome: Change From Baseline in Area of Allodynia - Cohort 2 - Week 4
Description: as for outcome 35
Time Frame: Baseline to Week 4
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: Square Centimeters (cm^2)
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 58 | 59
Square Centimeters (cm^2) | -54.33 [-72.041 to -13.677] | -69.39 [-116.234 to -45.112]

41. Secondary Outcome: Change From Baseline in Area of Allodynia - Cohort 2 - Week 8
Description: as for outcome 35
Time Frame: Baseline to Week 8
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: Square Centimeters (cm^2)
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 53 | 57
Square Centimeters (cm^2) | -78.78 [-99.958 to -43.748] | -75.58 [-113.401 to -50.634]

42. Secondary Outcome: Change From Baseline in Area of Allodynia - Cohort 2 - Week 12
Description: as for outcome 35
Time Frame: Baseline to Week 12
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: Square Centimeters (cm^2)
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 54 | 57
Square Centimeters (cm^2) | -77.98 [-99.148 to -36.515] | -79.99 [-129.775 to -49.428]

43. Secondary Outcome: Change From Baseline in Evoked Pain Score in the Area of Allodynia Cohort 1 - Week 2
Description: Assessment of evoked pain were conducted by a qualified and trained investigator or designee (eg, physician, physician's assistant, nurse practitioner, and nurse). Evoked pain was scored using a visual analog scale (VAS; 0 to100 mm scale with anchors of 0 = No pain and 100 = Worst pain imaginable). The patient was asked to use the VAS to rate the unpleasantness of 3 brush strokes within the center of the area of allodynia and pain.
Time Frame: Baseline to Week 2
Population: as for outcome 27
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 48 | 21 | 50
units on a scale | -17.4 [-25.67 to -10.68] | -21.2 [-30.01 to -10.09] | -15.3 [-22.76 to -7.32]

44. Secondary Outcome: Change From Baseline in Evoked Pain Score in the Area of Allodynia Cohort 1 - Week 4
Description: as for outcome 43
Time Frame: Baseline to Week 4
Population: as for outcome 27
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 50 | 25 | 51
units on a scale | -21.9 [-29.67 to -15.57] | -20.5 [-28.34 to -11.34] | -12.3 [-19.02 to -5.01]

45. Secondary Outcome: Change From Baseline in Evoked Pain Score in the Area of Allodynia Cohort 1 - Week 8
Description: as for outcome 43
Time Frame: Baseline to Week 8
Population: as for outcome 27
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 51 | 22 | 49
units on a scale | -22.7 [-31.18 to -15.80] | -24.8 [-34.73 to -14.45] | -19.4 [-27.27 to -10.15]

46. Secondary Outcome: Change From Baseline in Evoked Pain Score in the Area of Allodynia Cohort 1 - Week 12
Description: as for outcome 43
Time Frame: Baseline to Week 12
Population: as for outcome 27
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Number analyzed (Participants) | 51 | 23 | 46
units on a scale | -19.2 [-27.51 to -12.14] | -21.6 [-33.46 to -9.41] | -21.5 [-28.99 to -12.79]

47. Secondary Outcome: Change From Baseline in Evoked Pain Score in the Area of Allodynia - Cohort 2 - Week 2
Description: as for outcome 43
Time Frame: Baseline to Week 2
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 53 | 55
units on a scale | -19.0 [-26.102 to -11.030] | -16.2 [-23.400 to -9.691]

48. Secondary Outcome: Change From Baseline in Evoked Pain Score in the Area of Allodynia - Cohort 2 - Week 4
Description: as for outcome 43
Time Frame: Baseline to Week 4
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 52 | 55
units on a scale | -20.6 [-27.941 to -10.867] | -20.5 [-29.487 to -13.640]

49. Secondary Outcome: Change From Baseline in Evoked Pain Score in the Area of Allodynia - Cohort 2 - Week 8
Description: as for outcome 43
Time Frame: Baseline to Week 8
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 48 | 52
units on a scale | -28.7 [-35.924 to -21.285] | -19.7 [-27.721 to -11.895]

50. Secondary Outcome: Change From Baseline in Evoked Pain Score in the Area of Allodynia - Cohort 2 - Week 12
Description: as for outcome 43
Time Frame: Baseline to Week 12
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | AGN 214868 130µg | Placebo
Number analyzed (Participants) | 47 | 51
units on a scale | -26.9 [-37.750 to -16.548] | -19.1 [-26.996 to -10.612]

ADVERSE EVENTS:
Arm/Group | AGN 214868 130µg | AGN 214868 65µg | AGN 214868 32.5µg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/64 | 8/63 | 2/30 | 10/123
Other Adverse Events (participants affected / at risk) | 15/64 | 15/63 | 8/30 | 30/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AGN 214868 130µg (N=64) | AGN 214868 65µg (N=63) | AGN 214868 32.5µg (N=30) | Placebo (N=123)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Urethral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint crepitation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Thalamic infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AGN 214868 130µg (N=64) | AGN 214868 65µg (N=63) | AGN 214868 32.5µg (N=30) | Placebo (N=123)
Injection site pain (General disorders) | 6 | 1 | 0 | 6
Upper respiratory tract infection (Infections and infestations) | 4 | 5 | 1 | 8
Nasopharyngitis (Infections and infestations) | 3 | 5 | 2 | 9
Dizziness (Nervous system disorders) | 1 | 2 | 3 | 2
Urinary tract infection (Infections and infestations) | 1 | 2 | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other